CLINICAL TRIAL: NCT05396521
Title: Utilizing Blood Flow Restriction Therapy Following ORIF Treated Distal Radius Fractures
Brief Title: BFR Therapy Following DRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Peter J Apel, Orthopaedic surgeon, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-21-1514
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2023-05

CONDITIONS: Distal Radius Fracture
Keywords: Blood Flow Restriction
MeSH Terms: conditions — Wrist Fractures | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care Physical Therapy
- Blood Flow Restriction Supplemented (Experimental)
  Interventions: Other: Blood Flow Restriction

INTERVENTIONS:
Other: Blood Flow Restriction — Group 2 (experimental) will receive standard of care physical therapy to be done with blood flow restriction therapy (BFR). This method includes standard of care physical therapy while occluding blood flow.
  Arms: Blood Flow Restriction Supplemented
Other: Standard of Care Physical Therapy — Group 1 (Control) will receive standard of care physical therapy.
  Arms: Standard of Care

SUMMARY:
This study's goal is to evaluate whether blood flow restriction supplemented therapy is a superior therapy compared to traditional standard of care while recovering from a surgery that repairs distal radius fractures. In order to measure this, subjects will be randomly assigned to either the traditional therapy group (with standard of care) or a blood flow restriction supplemented therapy group. All patients involved in this study will have had a distal radius fracture that is repaired with a technique called volar plating and the procedure will be done via an open technique. All subjects will be asked to fill out questionnaires that assess their pain and wrist functionality throughout the course of the study. These measurements will help understand whether the supplemented therapy is effective at reducing pain and improving functionality for patients who are recovering from this injury.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients undergoing distal radius fracture open reduction internal fixation using volar plating (CPT 25607, 25608, and 25609)
* Age 50 - 75
* Fall onto outstretched hand injury

Exclusion Criteria:

* High energy mechanism

  * Fall from an elevated position greater than 12 inches
  * Motor vehicle collision
  * Any activity involving a powered vehicle (scooter, car, truck, ATV, motorcycle, tractor, etc.)
* any concomitant injury to the affected limb
* Bilateral distal radius fracture
* Revision procedures
* Worker's compensation status
* Non-English speaking
* No Internet Access
* Inability to provide informed consent
* Patients with known lymphovascular disorders, including peripheral arterial disease (PAD), prior deep vein thrombosis (DVT) or chronic lymphedema
* Patients with known genetic or other hypercoagulability disorders including those on long-term anticoagulation or anti-platelet therapy (other than prophylactic aspirin)
* Uncontrolled hypertension
* Patients with dialysis catheters or AV fistula
* Any other medical condition that affects the risk profile of the patient or that affects the normal physiologic function of the circulatory system of the extremities, based on sole discretion and medical judgement of the Primary Investigator

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain interference SF V1.1 | 3 months
PRWE | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corsino CB, Reeves RA, Sieg RN. Distal Radius Fractures. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536916/ PMID 30725601
- [Background] Pope D, Tang P. Carpal Tunnel Syndrome and Distal Radius Fractures. Hand Clin. 2018 Feb;34(1):27-32. doi: 10.1016/j.hcl.2017.09.003. PMID 29169594
- [Background] Kooner P, Grewal R. Is Therapy Needed After Distal Radius Fracture Treatment, What Is the Evidence? Hand Clin. 2021 May;37(2):309-314. doi: 10.1016/j.hcl.2021.02.012. PMID 33892883
- [Background] Shinohara M, Kouzaki M, Yoshihisa T, Fukunaga T. Efficacy of tourniquet ischemia for strength training with low resistance. Eur J Appl Physiol Occup Physiol. 1998;77(1-2):189-91. doi: 10.1007/s004210050319. PMID 9459541
- [Background] Takarada Y, Takazawa H, Ishii N. Applications of vascular occlusion diminish disuse atrophy of knee extensor muscles. Med Sci Sports Exerc. 2000 Dec;32(12):2035-9. doi: 10.1097/00005768-200012000-00011. PMID 11128848
- [Background] Gundermann DM, Walker DK, Reidy PT, Borack MS, Dickinson JM, Volpi E, Rasmussen BB. Activation of mTORC1 signaling and protein synthesis in human muscle following blood flow restriction exercise is inhibited by rapamycin. Am J Physiol Endocrinol Metab. 2014 May 15;306(10):E1198-204. doi: 10.1152/ajpendo.00600.2013. Epub 2014 Apr 1. PMID 24691032
- [Background] Loenneke JP, Fahs CA, Wilson JM, Bemben MG. Blood flow restriction: the metabolite/volume threshold theory. Med Hypotheses. 2011 Nov;77(5):748-52. doi: 10.1016/j.mehy.2011.07.029. Epub 2011 Aug 12. PMID 21840132
- [Background] Fry CS, Rasmussen BB. Skeletal muscle protein balance and metabolism in the elderly. Curr Aging Sci. 2011 Dec;4(3):260-8. doi: 10.2174/1874609811104030260. PMID 21529326
- [Background] Nielsen JL, Aagaard P, Bech RD, Nygaard T, Hvid LG, Wernbom M, Suetta C, Frandsen U. Proliferation of myogenic stem cells in human skeletal muscle in response to low-load resistance training with blood flow restriction. J Physiol. 2012 Sep 1;590(17):4351-61. doi: 10.1113/jphysiol.2012.237008. Epub 2012 Jul 16. PMID 22802591
- [Background] Moritani T, Sherman WM, Shibata M, Matsumoto T, Shinohara M. Oxygen availability and motor unit activity in humans. Eur J Appl Physiol Occup Physiol. 1992;64(6):552-6. doi: 10.1007/BF00843767. PMID 1618195
- [Background] Wernbom M, Augustsson J, Raastad T. Ischemic strength training: a low-load alternative to heavy resistance exercise? Scand J Med Sci Sports. 2008 Aug;18(4):401-16. doi: 10.1111/j.1600-0838.2008.00788.x. Epub 2008 May 3. PMID 18466185
- [Background] Shakeel R, Khan AA, Ayyub A, Masood Z. Impact of strengthening exercises with and without blood flow restriction on quadriceps of knee osteoarthritis patients. J Pak Med Assoc. 2021 Sep;71(9):2173-2176. doi: 10.47391/JPMA.377. PMID 34580509
- [Background] Cheema AS, O'Brien PJ, Broekhuyse HM, Lefaivre KA. Measuring Outcomes Over Time in Distal Radius Fractures: A Comparison of Generic, Upper Extremity-Specific and Wrist-Specific Outcome Measures. J Hand Surg Glob Online. 2020 Aug 14;2(5):272-276. doi: 10.1016/j.jhsg.2020.06.006. eCollection 2020 Sep. PMID 35415515
- [Background] MacDermid JC. The PRWE/PRWHE update. J Hand Ther. 2019 Apr-Jun;32(2):292-294. doi: 10.1016/j.jht.2019.01.001. Epub 2019 Mar 25. No abstract available. PMID 30922707